CLINICAL TRIAL: NCT06937229
Title: A Phase 3, Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of KarXT + KarX-EC for the Treatment of Agitation Associated With Alzheimer's Disease (ADAGIO-3)
Brief Title: A Study to Evaluate the Long-term Efficacy and Safety of KarXT + KarX-EC for Agitation in Alzheimer's Disease (ADAGIO-3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0025; 2024-519994-20 (Other: EU CTR); U1111-1316-3903 (Other: WHO)
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Agitation
Keywords: Agitation; Alzheimer disease; KarXT; KarX-EC
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation | interventions — xanomeline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT+KarX-EC (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: Xanomeline and Trospium Chloride capsule, BMS-986510
Drug: KarX-EC — Specified dose on specified days
  Other Names: Xanomeline enteric capsules, BMS-986519

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of combined formulation of xanomeline tartrate/trospium chloride in an immediate release (IR) capsule (KarXT) and xanomeline enteric capsules (KarX-EC) in participants with agitation associated with Alzheimer's Disease who completed the parent studies CN012-0023 or CN012-0024.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed study CN012-0023 or CN012-0024 per protocol.
* Participants must have one identified caregiver who should have sufficient contact (approximately 10 hours a week or more).

Exclusion Criteria:

* Participants must not have clinically significant cardiovascular (eg, untreated or unstable hypertension, clinically significant tachycardia), pulmonary, renal, hematologic, GI, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-06-22 (Estimated); Study Completion 2029-07-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately Week 30

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately Week 30
Number of Participants With Serious AEs (SAEs) | Up to approximately Week 30
Number of Participants With TEAEs Leading to Study Withdrawal | Up to approximately Week 30
Number of Participants With TEAEs Leading to Death | Up to approximately Week 30
Number of Participants with Adverse Events of Special Interest (AESI) | Up to approximately Week 30
Change From Baseline in Barnes Akathisia Rating Scale (BARS) | Up to approximately Week 26
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) | Up to approximately Week 26
Change From Baseline in Body Weight | Up to approximately Week 26
Change From Baseline in Body Mass Index (BMI) | Up to approximately Week 26
Number of Participants With Clinically Significant Changes in Orthostatic Vital Sign: Heart Rate (HR) | Up to approximately Week 30
  This includes measuring of HR, both supine and standing or seated and upon standing after 2 minutes.
Number of Participants With Clinically Significant Changes in Orthostatic Vital Sign: Blood Pressure (BP) | Up to approximately Week 30
  This includes measuring of systolic and diastolic BP, both supine and standing or seated and upon standing after 2 minutes.
Number of Participants With Clinically Significant Changes in Laboratory Evaluations | Up to approximately Week 30
Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) | Up to approximately Week 26
Number of Participants With Suicidal Ideations as Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately Week 30
Number of Participants With Cognitive Impairment as Assessed by Mini-mental State Examination (MMSE) | Up to approximately Week 26
Number of Participants With Cognitive Impairment as Assessed by 13-item Variation of ADAS-Cog Scale (ADAS-Cog-13) | Up to approximately Week 26
Change From Baseline in the Severity of Benign Prostatic Hyperplasia as Assessed by International Prostate Symptom Score (IPSS) | Up to approximately Week 26
  This analysis is done in male participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (244):
- United States (49):
  - Local Institution - 2609, Chandler, Arizona
  - Imaging Endpoints, Scottsdale, Arizona
  - Local Institution - 1657, Anaheim, California
  - Local Institution - 2620, Canoga Park, California
  - Local Institution - 1637, La Jolla, California
  - Local Institution - 2625, Long Beach, California
  - Local Institution - 2607, Long Beach, California
  - Local Institution - 2642, Long Beach, California
  - Local Institution - 2613, Pasadena, California
  - Local Institution - 1662, Pomona, California
  - Local Institution - 2614, San Diego, California
  - Local Institution - 1651, Walnut Creek, California
  - Local Institution - 2602, Bonita Springs, Florida
  - Local Institution - 2626, Hialeah, Florida
  - Local Institution - 1602, Miami, Florida
  - Local Institution - 1618, Miami, Florida
  - Local Institution - 1609, Miami, Florida
  - Nuovida Research Center, Miami, Florida
  - Local Institution - 1635, Orlando, Florida
  - Local Institution - 1612, Port Orange, Florida
  - Local Institution - 2621, Tampa, Florida
  - Local Institution - 1636, Gaithersburg, Maryland
  - Local Institution - 1638, Newton, Massachusetts
  - Local Institution - 2615, Worcester, Massachusetts
  - Local Institution - 2618, Ann Arbor, Michigan
  - Local Institution - 1620, Troy, Michigan
  - Local Institution - 2256, Saint Paul, Minnesota
  - Local Institution - 2629, Hattiesburg, Mississippi
  - Local Institution - 2628, Las Vegas, Nevada
  - Local Institution - 1649, Las Vegas, Nevada
  - Local Institution - 1647, West Long Branch, New Jersey
  - Local Institution - 1656, New Windsor, New York
  - Local Institution - 2619, Staten Island, New York
  - Local Institution - 1658, Woodmere, New York
  - Local Institution - 1601, Monroe, North Carolina
  - Local Institution - 2608, Morehead City, North Carolina
  - Local Institution - 2617, Blue Ash, Ohio
  - Local Institution - 1640, Tulsa, Oklahoma
  - Local Institution - 1653, Columbia, South Carolina
  - Epic Medical Research, LLC - Carrolton, Carrollton, Texas
  - Local Institution - 2605, Cypress, Texas
  - Local Institution - 1643, El Paso, Texas
  - Local Institution - 2622, Mesquite, Texas
  - Local Institution - 2623, San Antonio, Texas
  - Pantheon Clinical Research, LLC, Bountiful, Utah
  - Local Institution - 1646, Bennington, Vermont
  - Local Institution - 1644, Seattle, Washington
  - Local Institution - 1654, Spokane, Washington
  - Local Institution - 2610, Milwaukee, Wisconsin
- Argentina (14):
  - Local Institution - 2005, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 1001, La Plata, Buenos Aires
  - Local Institution - 1002, Mar del Plata, Buenos Aires
  - Local Institution - 2006, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 1006, Rosario, Santa Fe Province
  - Local Institution - 2004, Buenos Aires
  - Local Institution - 1003, Buenos Aires
  - Local Institution - 1004, Córdoba
  - Local Institution - 2000, Córdoba
  - Local Institution - 2002, Córdoba
  - Local Institution - 1005, Córdoba
  - Local Institution - 1000, Córdoba
  - Local Institution - 2003, Córdoba
  - Local Institution - 2001, Mendoza
- Brazil (9):
  - Local Institution - 1051, Brasília, Federal District
  - Local Institution - 1053, Curitiba, Paraná
  - Local Institution - 1052, Curitiba, Paraná
  - Local Institution - 1058, Porto Alegre, Rio Grande do Sul
  - Local Institution - 1054, Porto Alegre, Rio Grande do Sul
  - Local Institution - 1057, Campinas, São Paulo
  - Local Institution - 1056, São Paulo, São Paulo
  - Local Institution - 1050, Rio de Janeiro
  - Local Institution - 1055, São Paulo
- Bulgaria (4):
  - Local Institution - 1100, Sofia, Sofia-Grad
  - Local Institution - 1101, Pleven
  - Local Institution - 1103, Razgrad
  - Local Institution - 1102, Varna
- Canada (5):
  - Local Institution - 1153, Hamilton, Ontario
  - Local Institution - 1155, London, Ontario
  - Local Institution - 1151, Toronto, Ontario
  - Local Institution - 1154, Toronto, Ontario
  - Local Institution - 1152, Whitby, Ontario
- Chile (5):
  - Local Institution - 2055, Viña del Mar, Región de Valparaíso
  - Local Institution - 2051, Santiago, Santiago Metropolitan
  - Local Institution - 2052, Santiago, Santiago Metropolitan
  - Local Institution - 2054, Vitacura, Santiago Metropolitan
  - Local Institution - 2053, Antofagasta
- Croatia (5):
  - Local Institution - 1553, Zagreb, City of Zagreb
  - Local Institution - 1554, Rijeka
  - Local Institution - 1551, Split
  - Local Institution - 1552, Varaždin
  - Local Institution - 1550, Zagreb
- Czechia (9):
  - Local Institution - 2107, Olomouc, Olomoucký kraj
  - Local Institution - 2100, Prague, Praha 6
  - Local Institution - 2106, Prague, Praha 8
  - Local Institution - 2103, Brno, South Moravian
  - Local Institution - 2101, Choceň
  - Local Institution - 2104, Pilsen
  - Local Institution - 2102, Prague
  - Local Institution - 2105, Prague
  - Local Institution - 2108, Rychnov nad Kněžnou
- France (7):
  - Local Institution - 2150, Toulouse, Haute-Garonne
  - Local Institution - 2151, Villeurbanne, Rhône
  - Local Institution - 2153, Lille
  - Local Institution - 2156, Limoges
  - Local Institution - 2157, Montpellier
  - Local Institution - 2152, Paris
  - Local Institution - 2155, Strasbourg
- Germany (4):
  - Local Institution - 2203, Erbach im Odenwald, Hesse
  - Local Institution - 2201, Düsseldorf
  - Local Institution - 2205, Halle
  - Local Institution - 2206, Westerstede
- Greece (9):
  - Local Institution - 1200, Pátrai, Achaḯa
  - Local Institution - 1205, Athens, Attica
  - Local Institution - 1202, Athens, Attica
  - Local Institution - 1203, Chaïdári, Attikí
  - Local Institution - 0027, Athens
  - Local Institution - 1206, Athens
  - Local Institution - 1207, Athens
  - Local Institution - 1201, Ioannina
  - Local Institution - 1204, Thessaloniki
- Hungary (7):
  - Local Institution - 2257, Kalocsa, Bács-Kiskun county
  - Local Institution - 2250, Győr, Győr-Moson-Sopron
  - Local Institution - 2254, Gyöngyös, Heves County
  - Local Institution - 2255, Budapest
  - Local Institution - 2251, Budapest
  - Local Institution - 2253, Budapest
  - Local Institution - 2252, Debrecen
- India (7):
  - Local Institution - 1251, Hyderabad, Andhra Pradesh
  - Local Institution - 1255, Ahmedabad, Gujarat
  - Local Institution - 1252, Hyderabad, Telangana
  - Local Institution - 1254, Varanasi, Uttar Pradesh
  - Local Institution - 1250, Kolkata, West Bengal
  - Local Institution - 1256, Delhi
  - Local Institution - 1253, New Delhi
- Israel (6):
  - Local Institution - 2302, Petch Tikva, IL
  - Local Institution - 2301, Jerusalem
  - Local Institution - 2303, Netanya
  - Local Institution - 2305, Ramat Gan
  - Local Institution - 2300, Ramat Gan
  - Local Institution - 2304, Rishon Le'Tzion
- Italy (8):
  - Local Institution - 2351, Napoli, Campania
  - Local Institution - 2354, Rome, Lazio
  - Local Institution - 2352, Rome, Lazio
  - Local Institution - 2353, Milan, Lombardy
  - Local Institution - 2350, Pisa, PI
  - Local Institution - 2356, Brescia
  - Local Institution - 2355, Isernia
  - Local Institution - 2357, Roma
- Japan (9):
  - Local Institution - 1301, Hadano, Kanagawa
  - Local Institution - 1307, Kawasaki, Kanagawa
  - Local Institution - 1304, Sakai, Osaka
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki-Gun Yoshinogari-Cho, Saga-ken
  - Rainbow and Sea Hospital, Karatsu-shi, Saga-ken
  - Local Institution - 1305, Bunkyo-ku, Tokyo
  - Kuramitsu Hospital, Fukuoka
  - Local Institution - 1306, Okayama
  - Local Institution - 1308, Shimotsuke-shi, Tochigi
- Mexico (9):
  - Local Institution - 1355, Saltillo, Coahuila
  - Local Institution - 1356, Guadajalara, Jalisco
  - Local Institution - 1350, Monterrey, Nuevo León
  - Local Institution - 1361, Mexico City
  - Local Institution - 1363, Mexico City
  - Local Institution - 1360, Mexico City
  - Local Institution - 1364, Monterrey
  - Local Institution - 1362, San Luis Potosí City
  - Local Institution - 1352, Tlalnepantla
- Poland (7):
  - Local Institution - 2450, Poznan, Greater Poland Voivodeship
  - Local Institution - 2454, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 2456, Chorzów
  - Local Institution - 2455, Katowice
  - Local Institution - 2451, Lublin
  - Local Institution - 2452, Lublin
  - Local Institution - 2453, Sochaczew
- Portugal (5):
  - Local Institution - 1401, Coimbra
  - Local Institution - 1402, Guimarães
  - Local Institution - 1404, Lisbon
  - Local Institution - 1403, Senhora da Hora
  - Local Institution - 1400, Torres Vedras
- Romania (13):
  - Local Institution - 1450, Bucharest, București
  - Local Institution - 1452, Bucharest, București
  - Local Institution - 1453, Bucharest, București
  - Local Institution - 1454, Bucharest, București
  - Local Institution - 1455, Bucharest, București
  - Local Institution - 1456, Bucharest, București
  - Local Institution - 1458, Bucharest, București
  - Local Institution - 1451, Bucharest
  - Local Institution - 1459, Bucharest
  - Local Institution - 1461, Constanța
  - Local Institution - 1457, Iași
  - Local Institution - 1460, Sanpetru /Brasov
  - Local Institution - 1462, Sibiu
- South Korea (10):
  - Local Institution - 2401, Incheon, Incheon Gwang'yeogsi
  - Local Institution - 2407, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 2403, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 2406, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 2400, Deagu, Taegu-Kwangyǒkshi
  - Local Institution - 2409, Incheon
  - Local Institution - 2402, Seoul
  - Local Institution - 2408, Seoul
  - Local Institution - 2405, Seoul
  - Local Institution - 2404, Seoul
- Spain (12):
  - Local Institution - 1510, Getxo, Bizkaia
  - Local Institution - 1509, Elche (alicante)
  - Local Institution - 1508, Madrid
  - Local Institution - 1505, Madrid
  - Local Institution - 0003, Málaga
  - Local Institution - 1502, Málaga
  - Local Institution - 1507, Pamplona
  - Local Institution - 1500, Salamanca
  - Local Institution - 1503, Seville
  - Local Institution - 1504, Terrassa
  - Local Institution - 1506, Valladolid
  - Local Institution - 1501, Zaragoza
- Taiwan (5):
  - Local Institution - 1753, Kaohsiung Niao Sung Dist, Kaohsiung
  - Local Institution - 1751, Tainan, Taiana
  - Local Institution - 1754, Taipei
  - Local Institution - 1750, Taipei
  - Local Institution - 1752, Taoyuan District
- Ukraine (16):
  - Local Institution - 2555, Smila, Cherkasy Oblast
  - Local Institution - 2554, Dnipro, Dnipropetrovsk Oblast
  - Local Institution - 2561, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Local Institution - 2559, Skarzhyntsi, Khmelnytskyi Oblast
  - Local Institution - 2556, Hlevakha, Kyiv Oblast
  - Local Institution - 2566, Hlevakha, Kyiv Oblast
  - Local Institution - 2553, Kyiv, Kyivska Oblast
  - Local Institution - 2552, Lviv, Lviv Oblast
  - Local Institution - 2558, Lviv, Lviv Oblast
  - Local Institution - 2569, Lviv, Lviv Oblast
  - Local Institution - 2567, Oleksandrivka, Odesa Oblast
  - Local Institution - 2557, Poltava, Poltava Oblast
  - Local Institution - 2551, Vinnytsia, Vinnytsia Oblast
  - Local Institution - 2550, Kropyvnytskyi
  - Local Institution - 2565, Kyiv
  - Local Institution - 2568, Odesa
- United Kingdom (10):
  - Local Institution - 2505, Preston, Lancashire
  - Local Institution - 2508, Chertsey, Surrey
  - Local Institution - 2502, Cambridge
  - Local Institution - 2501, London
  - Local Institution - 2500, London
  - Local Institution - 2510, Motherwell
  - Local Institution - 2507, Redruth
  - Local Institution - 2504, Sheffield
  - Local Institution - 2509, Stafford
  - Local Institution - 2503, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06937229.html